CLINICAL TRIAL: NCT00377468
Title: Low Dose Administration of Delta9-Tetrahydrocannabinol for the Prevention of Hyperalgesia and Chronic Pain in Patients With Acute Complex Regional Pain Syndrome (CRPS) of the Upper Limb
Brief Title: Effect of Delta-9-Tetrahydrocannabinol on the Prevention of Chronic Pain in Patients With Acute CRPS (ETIC-Study)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network on Neuropathic Pain (Network)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2310106; Eudra-CT: 2006-000439-85
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Complex Regional Pain Syndromes; CRPS
Keywords: THC; CRPS; Pain; Complex Regional Pain Syndrome; Neuropathic Pain; Chronic; Prevention
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain; Neuralgia; Bronchiolitis Obliterans Syndrome | interventions — Dronabinol

INTERVENTIONS:
Drug: Delta9-Tetrahydrocannabinol

SUMMARY:
The purpose of this study is to determine whether application of low dose Delta9-Tetrahydrocannabinol can prevent the development of chronic pain in patients with acute CRPS.

DETAILED DESCRIPTION:
Recent animal data suggest that the endocannabinoid system is a promising target in the prevention of chronic pain. It has been shown that the endocannabinoid system modifies excitatory and inhibitory currents in structures involved in the development of chronic pain such as the amygdala.

CRPS is a neuropathic pain condition, which is known to become chronic in a significant percentage. The study compares the effect of low dose Delta9-Tetrahydrocannabinol (90 days) and placebo in acute CRPS. All patients will receive a standard treatment consisting of drug therapy and physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of acute CRPS (time from inciting event less than 16 weeks) of the upper extremity
* No risk of dependency in a psychological assessment

Exclusion Criteria:

* History of alcohol or drug abuse
* Cardiac arrhythmias
* Acute or chronic renal failure
* ASA physical status classification III or higher
* Psychiatric disorders
* Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain at one year assessed with Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Changes in somatosensory phenotype at one year assessed with Quantitative Sensory Testing (QST)
Motor function of the affected extremity at one year assessed with a biometric evaluation
Changes in Health Related Quality of Life at one year assessed with SF-36
Changes in plasma endocannabinoid levels at 30, 60, 90 days and at one year

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz C Azad, MD;PhD, Principal Investigator — Department of Anesthesiology, Interdisciplinary Pain Clinic Grosshadern, University of Munich
Locations (1):
- Department of Anesthesiology, Interdisciplinary Pain Clinic Grosshadern, Universitiy of Munich, Munich, Germany

REFERENCES:
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Azad SC, Monory K, Marsicano G, Cravatt BF, Lutz B, Zieglgansberger W, Rammes G. Circuitry for associative plasticity in the amygdala involves endocannabinoid signaling. J Neurosci. 2004 Nov 3;24(44):9953-61. doi: 10.1523/JNEUROSCI.2134-04.2004. PMID 15525780
- [Background] Azad SC, Eder M, Marsicano G, Lutz B, Zieglgansberger W, Rammes G. Activation of the cannabinoid receptor type 1 decreases glutamatergic and GABAergic synaptic transmission in the lateral amygdala of the mouse. Learn Mem. 2003 Mar-Apr;10(2):116-28. doi: 10.1101/lm.53303. PMID 12663750